CLINICAL TRIAL: NCT00764985
Title: E-STOP Registry: A Registry for the Evaluation of Syncope,Its Diagnosis, Treatment, Outcome and Prognosis Using Our SELF-Pathway
Brief Title: Evaluation of Syncope,Its Diagnosis, Treatment, Outcome and Prognosis
Acronym: E-STOP
Status: Completed | Type: Observational
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Collaborators: Transoma Medical (Industry)
Responsible Party: Suneet Mittal, St. Luke's-Roosevelt Hospitals
Other Study IDs: ESTOP-08-024
Record Dates: First submitted 2008-10-01; First posted 2008-10-02 (Estimated); Last update posted 2010-07-02 (Estimated); Status verified 2010-07

CONDITIONS: Syncope
Keywords: Syncope; Pre-Syncope; Fainting
MeSH Terms: conditions — Syncope

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Syncope

SUMMARY:
The investigators want to look at how patients admitted after passing out (syncope) or nearly passing out (pre-syncope) do after going home and how many of them remain free of symptoms of syncope or pre-syncope.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (age 18 or older) admitted with syncope or near-syncope

Exclusion Criteria:

* Patients who do not speak/read the language of the consent form
* Prisoners
* Patients who are of altered mental status or had head trauma
* Refusal or inability to sign consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patietns admitted to the adult medicine service at St. Luke's-Roosevelt Hospital with diagnossi of syncope or near syncope
Sampling Method: Non-Probability Sample
Enrollment: 540 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- St. Luke's-Roosevelt Hospital Center, New York, New York, United States